CLINICAL TRIAL: NCT04993092
Title: Comparative Study on the Effects of Mulligan Mobilization Technique and Muscle Energy Technique on Pain and Range of Motion in Adhesive Capsulitis
Brief Title: Mulligan Mobilization Technique and Muscle Energy Technique on Pain and ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0115 Sumaira
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Adhesive Capsulitis
Keywords: Frozen shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mulligan mobilization technique (Experimental): Sustain Posterolateral glide with belt and then told Patient to move in following pattern (internal rotation, external rotation, abduction, wall sliding)
  Interventions: Other: mulligan mobilization technique
- muscle energy technique (Active Comparator): Post facilitation stretch Patient perform isometrics for 15 seconds then therapist rapidly move the shoulder to the end range
  Interventions: Other: muscle energy technique

INTERVENTIONS:
Other: muscle energy technique — Post facilitation stretch Patient perform isometrics for 15 seconds then therapist rapidly move the shoulder to the end range
  Arms: muscle energy technique
Other: mulligan mobilization technique — Sustain Posterolateral glide with belt and then told Patient to move in following pattern (internal rotation, external rotation, abduction, wall sliding)
  Arms: mulligan mobilization technique

SUMMARY:
this study will be a randomized clinical trial. This study will be conducted in Nishat Latif Hospital, Barath, Sialkot. A sample size of 22 patients will be taken. Patients will be divided into two groups by lottery method. Group A will be treated with mulligan mobilization technique and conventional physiotherapy with Transcutaneous electrical nerve stimulation and electrical heating pad. Group B will be treated with muscle energy technique and conventional treatment of Transcutaneous electrical nerve stimulation and electrical hot pack. Both groups will receive treatment for5 weeks,2 sessions in a week with baseline and 6 weeks treatment reading will be taken. The outcome measures Numeric pain rating scale, disabilities of the arm, shoulder and hand, Shoulder Pain and Disability Index . data will be analyzed by Statistical Package for the Social Sciences 25.

DETAILED DESCRIPTION:
Frozen shoulder, also known as adhesive capsulitis, is a condition characterized by stiffness and pain in your shoulder joint. A condition in which a person has severe limitation of the range of motion of the shoulder due to scarring around the shoulder joint. Adhesive capsulitis is an unwanted consequence of rotator cuff disease that involves damage to the rotator cuff. Muscle energy technique involves careful positioning of an area of the body by the physical therapist. After positioning, you will be asked to contract the muscle or resist a movement done by the physical therapist. This will be followed by a stretch to lengthen the same or opposite muscle group.

This will be followed by a stretch to lengthen the same or opposite muscle group. Mulligan's technique "combines the sustained application of manual gliding force to a joint, with the aim of repositioning bone positional faults while enabling concurrent physiological (osteo-kinematic) motion of the joint. Essentially, this means repositioning a joint to enable proper motion while taking that joint through pain-free passive and active range of motion (ROM).

Mulligan Manual Therapy can be used to help treat a variety of injuries and pain including neck pain, back pain and upper and lower extremity injuries. Designed to reduce pain and improve the patient's range of motion the Mulligan technique involves Natural Apophyseal Glides (NAGS), Sustained Natural Apophyseal Glides (SNAGS) and Mobilization with Movement (MWM) for the treatment of musculoskeletal injuries.

The American Academy of Orthopedic Surgeons describe three stages: Freezing, or painful stage: Pain increases gradually, making shoulder motion harder and harder. Pain tends to be worse at night. Frozen: Pain does not worsen, and it may decrease at this stage. The shoulder remains stiff. Thawing: Movement gets easier and may eventually return to normal. Signs and symptoms typically begin gradually, worsen over time and then resolve, usually within one to three years.

ELIGIBILITY:
Inclusion Criteria:

* Pain in shoulder for at least 3 months
* Unilateral frozen shoulder of stage 3 and 4
* Capsular pattern i.e. (lateral rotation, Abduction, Medial rotation)

Exclusion Criteria:

* Secondary capsulitis
* Shoulder injury such as proximal humerus fracture.
* History of Neurological deficit i.e. cervical stenosis, myelopathy.
* Prolong immobilization due to cardiothoracic surgery, neurosurgery.
* Shoulder surgical history such as shoulder arthroplasty.
* History of other pathological condition of shoulders i.e. Impingement syndrome, rotator cuff tear or any shoulder injury

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
The Quick Disabilities of the Arm, Shoulder and Hand | 4th week
  The Quick Disabilities of the Arm, Shoulder and Hand only contains subset of 11 items. it is a self-reported questionnaire in which the response options are presented as 5-point Likert scales.
  At least 10 of the 11 items must be completed for a score to be calculated The scores range from 0 (no disability) to 100 (most severe disability).
The Shoulder Pain and Disability Index | 4th week
  it is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with activity of daily living requiring the use of the upper extremities. The pain subscale is a composite measure and has 5-items and the Disability subscale is a composite measure and has 8-items.
  Total pain score (which is composite measure): / 50 x 100 = % (Note: If a person does not answer all questions divide by the total possible score, eg. if 1 question missed divide by 40)
  Total disability score (which is composite measure): / 80 x 100 = % (Note: If a person does not answer all questions divide by the total possible score, eg. if 1 question missed divide by 70)
  Total Shoulder Pain and Disability score: / 130 x 100 = % (Note: If a person does not answer all questions divide by the total possible score, eg. if 1 question missed divide by 120)
  The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Goniometry | 4th week
  To measure Range of Motion at Shoulder joint.

SECONDARY OUTCOMES:
Numeric pain rating scale | 4th week
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator
Locations (1):
- Sumaira Nawaz, Sialkot, Sialkot,Punjab,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodridge JP. Muscle energy technique: definition, explanation, methods of procedure. J Am Osteopath Assoc. 1981 Dec;81(4):249-54. No abstract available. PMID 7319853
- [Background] Campbell SM, Winkelmann RR, Walkowski S. Osteopathic manipulative treatment: novel application to dermatological disease. J Clin Aesthet Dermatol. 2012 Oct;5(10):24-32. PMID 23125887
- [Background] Jain TK, Sharma NK. The effectiveness of physiotherapeutic interventions in treatment of frozen shoulder/adhesive capsulitis: a systematic review. J Back Musculoskelet Rehabil. 2014;27(3):247-73. doi: 10.3233/BMR-130443. PMID 24284277
- [Background] Yeganeh Lari A, Okhovatian F, Naimi Ss, Baghban AA. The effect of the combination of dry needling and MET on latent trigger point upper trapezius in females. Man Ther. 2016 Feb;21:204-9. doi: 10.1016/j.math.2015.08.004. Epub 2015 Aug 14. PMID 26304789
- [Background] Jones S, Hanchard N, Hamilton S, Rangan A. A qualitative study of patients' perceptions and priorities when living with primary frozen shoulder. BMJ Open. 2013 Sep 26;3(9):e003452. doi: 10.1136/bmjopen-2013-003452. PMID 24078753
- [Background] Solomonow M, Krogsgaard M. Sensorimotor control of knee stability. A review. Scand J Med Sci Sports. 2001 Apr;11(2):64-80. doi: 10.1034/j.1600-0838.2001.011002064.x. PMID 11252464
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Doner G, Guven Z, Atalay A, Celiker R. Evalution of Mulligan's technique for adhesive capsulitis of the shoulder. J Rehabil Med. 2013 Jan;45(1):87-91. doi: 10.2340/16501977-1064. PMID 23037929
- [Background] Nicholson GG. The effects of passive joint mobilization on pain and hypomobility associated with adhesive capsulitis of the shoulder. J Orthop Sports Phys Ther. 1985;6(4):238-46. doi: 10.2519/jospt.1985.6.4.238. PMID 18802309